CLINICAL TRIAL: NCT01352442
Title: A Prospective Multicenter Clinical Trial to Evaluate the Safety and Effectiveness of the AcuFocus Corneal Inlay ACI 7000PDT Implanted Intrastromally for Modified Monovision in Presbyopic Subjects
Brief Title: Safety and Effectiveness of the AcuFocus Corneal Inlay ACI7000PDT in Presbyopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACU-P10-020B
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Presbyopia
Keywords: Presbyopia; Accommodation; Near visual acuity; LASIK
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AcuFocus Corneal Inlay (Experimental): The AcuFocus Corneal Inlay ACI 7000PDT, which is a small medical device, will be surgically implanted in one eye of each subject.
  Interventions: Device: AcuFocus Corneal Inlay ACI 7000PDT

INTERVENTIONS:
Device: AcuFocus Corneal Inlay ACI 7000PDT — corneal inlay
  Other Names: AcuFocus KAMRA inlay

SUMMARY:
The purpose of this study is to determine if the AcuFocus Corneal Inlay ACI 7000PDT will provide an effective method of for the correction of presbyopia in patients who have normal distance vision but need correction such as glasses or contact lenses to see clearly at near.

DETAILED DESCRIPTION:
The design and mechanism of action of the AcuFocus™ Corneal Inlay (ACI 7000PDT) is based on the well-established concept of small-aperture optics. In cameras, depth of focus is controlled by reducing the aperture through which light enters; the smaller the aperture, the greater the depth of focus. This concept also applies to the human eye. In the eye of an emmetropic presbyope, the natural lens cannot fully accommodate to focus the light rays from a near object onto a single point on the retina. Thus, a point object is imaged as a blur circle on the retina, and images of extended objects are degraded as well. If an opaque disc with a small aperture in the center is placed in front of the eye, the peripheral rays will be obscured while the central rays pass unaffected. Since peripheral rays enter the eye at a larger angle, they create a larger blur circle at the retinal image plane. Eliminating these peripheral rays reduces the size of the blur circle, improving image resolution.

When the inlay is implanted in one eye, the increased depth of focus provides near and intermediate visual acuity while having a minimal effect on distance acuity. Under binocular conditions, the effect of having an inlay eye with a range of vision from distance to near combined with the uncorrected vision in the fellow presbyopic eye, which will essentially have good distance acuity with reduced near acuity, is similar to the contact lens modality known as "modified monovision."

The ACI is expected to provide presbyopic patients with improvement in near and intermediate vision.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign and be given a copy of the written Informed Consent form.
2. Subjects must be emmetropes needing a magnitude of +1.00D to +2.50D of reading add.
3. Subjects must have distance corrected near visual acuity worse than 20/40 and better than 20/100 in the eye to be implanted.
4. Subjects must have distance visual acuity correctable to at least 20/20 in both eyes.
5. Subjects must have a preoperative spherical equivalent of plano defined as Plano to -0.75D with no more than 0.75D of refractive cylinder as determined by cycloplegic refraction in the eye to be implanted.
6. Subjects must have a stable refraction twelve months prior to ACI implantation: i.e. MRSE within 0.50D over prior twelve months as determined by subject history.
7. Subjects who are soft contact lens wearers must discontinue their contact lenses for at least one week prior to ACI pre-operative examination.
8. Subjects must have a minimum central corneal thickness of ≥ 500 microns in the eye to be implanted.
9. Subjects must have a corneal power of ≥ 41.00D and ≤ 47.00D in all meridians in the eye to be implanted.
10. Subjects must be ≥ 45 years and ≤ 60 years of age at the time of subject eligibility visit.
11. Subjects must have an endothelial cell count ≥ 2000 cells/mm2 in the eye to be implanted.
12. Subjects must be willing and able to return for scheduled follow-up examinations for 12 months after surgery.
13. Subjects must demonstrate tolerance to monovision blur in the eye to be implanted as determined by loose lens blur tolerance or monovision contact lens trial.

Exclusion Criteria:

1. Subjects with a difference of >1.00D between the spherical equivalent manifest refraction and the spherical equivalent cycloplegic refraction.
2. Subjects with anterior segment pathology, including cataracts, in the eye to be implanted.
3. Subjects with residual, recurrent, active ocular or uncontrolled eyelid disease, or any corneal abnormality (including endothelial dystrophy, guttata, recurrent corneal erosion, etc.) in the eye to be implanted.
4. Subjects with ophthalmoscopic or topographic signs of keratoconus (or keratoconus suspect) or keratoectasia in the eye to be implanted.
5. Subjects with dry eye as determined by objective testing; anesthetized Schirmer's test result <10 mm or a tear break-up time (TBUT) less than 10 seconds are excluded.
6. Subjects taking chronic systemic medications known to exacerbate or induce moderate to severe dry eye in so far as measures of TBUT and Schirmers are decreased or borderline per Exclusion Criterion #5. Subjects taking the following classes of medications should be evaluated: anti-depressants, anti-histamines, beta-blockers, phenothiazines, atropine and atropine derivatives, oral contraceptives, anxiolytics, diuretics, anti-cholinergics, and anti-arrhythmics.
7. Subjects with distorted or unclear corneal mires on topography maps of the eye to be implanted.
8. Subjects with macular degeneration, retinal detachment, or any other fundus pathology that would prevent an acceptable visual outcome in the eye to be implanted.
9. Subjects who have worn RGP or PMMA contact lenses within the last 6 months.
10. Subjects who have undergone previous intraocular or corneal surgery, including PRK, LASIK, CK, LASEK, and cataract surgery in the eye to be implanted.
11. Subjects with a history of herpes zoster or herpes simplex keratitis.
12. Subjects who have a history of steroid-responsive rise in intraocular pressure, preoperative IOP > 21 mmHg, glaucoma, ocular hypertension, or are glaucoma suspects.
13. Subjects with an abnormal threshold visual field.
14. Subjects with a history of diagnosed diabetes, diagnosed autoimmune disease, connective tissue disease, or clinically significant atopic syndrome.
15. Subjects on chronic systemic corticosteroids or other immunosuppressive therapy that may affect wound healing, and any immunocompromised subjects.
16. Subjects who are using ophthalmic medication(s) other than artificial tears for treatment of any ocular pathology including ocular allergy.
17. Subjects using systemic medications with significant ocular side effects.
18. Subjects who are pregnant, lactating, or of child-bearing potential and not practicing a medically approved method of birth control.
19. Subjects with known sensitivity to planned study concomitant medications.
20. Subjects who are participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Binder, MD, Study Director
Locations (11):
- Vision Eye Institute, Bondi Junction, New South Wales, Australia
- Univ. Klinik fur Agugenheilkunde und Optometrie, Paracelsus Medzinishe Privatuniversitat Salzburg, Salzburg, Austria
- Fondation Rothchild, Paris, France
- Shinagawa Lasik Center, Tokyo, Japan
- Maastricht University Medical Center, Maastricht, Netherlands
- New Zealand (2):
  - The Fendalton Eye Clinic, Fendalton, Christchurch
  - Auckland Eye, Auckland
- Asian Eye Institute, Makati City, Philippines
- Singapore National Eye Centre, Singapore, Singapore
- CEIC Vissum Corporación Oftalmológica, Alicante, Spain
- Beyoğlu Goz Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://www.acufocus.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AcuFocus Corneal Inlay
Started | 151
Completed | 139
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | AcuFocus Corneal Inlay
Number analyzed (Participants) | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 151
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 80
Region of Enrollment [Number; unit: participants]
  Austria | 9
  Japan | 9
  Singapore | 8
  Philippines | 26
  Turkey | 36
  New Zealand | 16
  Australia | 26
  Spain | 3
  Netherlands | 6
  France | 12

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Near Visual Acuity 20/32 or Better
Time Frame: 12 months
Measure: Number; unit: percentage of subjects
Arm/Group | AcuFocus Corneal Inlay
Number analyzed (Participants) | 139
percentage of subjects | 73.8

2. Secondary Outcome: Subjective Rating of Near Visual Acuity at 12 Months as Measured by Subjective Questionnaire
Description: Mean subjective rating via questionnaire on 1 to 7 rating scale (1= very dissatisfied and 7 = very satisfied).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | AcuFocus Corneal Inlay
Number analyzed (Participants) | 139
Scores on a scale | 5.4 [2.3 to 8.5]

ADVERSE EVENTS:
Time Frame: 3 months, 6 months, 1 year, 2 years, 3 years
Arm/Group | AcuFocus Corneal Inlay
Serious Adverse Events (participants affected / at risk) | 7/151
Other Adverse Events (participants affected / at risk) | 34/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AcuFocus Corneal Inlay (N=151)
Complete division of left Achilles tendon (Musculoskeletal and connective tissue disorders) | 1 — All Serious Adverse Events reported in this study were not related to the eye.
Brain and Lung cancer requiring extended hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — All Serious Adverse Events reported in this study were not related to the eye.
Hospitalization for investigation of bladder. Suspected cancer. Planned event. (Investigations) | 1 — All Serious Adverse Events reported in this study were not related to the eye.
Hospitalization for laser treatment of bladder cancer. Planned event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — All Serious Adverse Events reported in this study were not related to the eye.
Hospitalisation for Systemic Cellulitis (Skin and subcutaneous tissue disorders) | 1 — All Serious Adverse Events reported in this study were not related to the eye.
Hospitalization for Atrial Fibrilation (Cardiac disorders) | 1 — All Serious Adverse Events reported in this study were not related to the eye.
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — All Serious Adverse Events reported in this study were not related to the eye.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AcuFocus Corneal Inlay (N=151)
Corneal Edema with grade of greater than or equal to 2+ (at one month or later) (Eye disorders) | 2
Epithelial Ingrowth (Eye disorders) | 2
Intraocular pressure (Eye disorders) | 7 — Intraocular pressure increase greater than 10 mmHg above baseline or Intraocular pressure greater than 25 mmHg (with clinical findings)
Allergic reaction to study medication (lids) (Eye disorders) | 1
Blepharitis (Eye disorders) | 1
AcuFocus Corneal Inlay re-centration or replacement (Eye disorders) | 9
Dry eye (Eye disorders) | 1
Decrease in Best Corrected Distance Visual Acuity greater than 2 lines at Month 3 or later (Eye disorders) | 6
Bone fracture (Injury, poisoning and procedural complications) | 2
Adenoviral Conjunctivitis (Eye disorders) | 1
Atrial Fibrilation (Cardiac disorders) | 1
Flap complication (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No